CLINICAL TRIAL: NCT00863148
Title: A Phase II Open-label, Multicenter, Non Randomized Study Evaluating the Efficacy and the Safety of Clofarabine in Combination With IV Busulfan and Thymoglobulin (CBT) as a Reduced Intensity Conditioning Regimen Prior to Allogeneic Stem Cell Transplantation in Adult Patients With High-risk AML, MDS or ALL.
Brief Title: Allogeneic Stem Cell Transplant With Clofarabine, Busulfan and Antithymocyte Globulin (ATG) for Adult Patients With High-risk Acute Myeloid Leukemia/Myelodysplastic Syndromes (AML/MDS) or Acute Lymphoblastic Leukemia (ALL)
Acronym: Cloric
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/08/07-J
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: MDS; AML; ALL; BAL
Keywords: MDS; AML; ALL; RIC; clofarabine; allo-HSCT; high-risk MDS/AML
MeSH Terms: interventions — Clofarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Clofarabine in combination with IV busulfan and ATG — A conservative approach has been used for the determination of the dose due to the high risk studied population, e.g., decrease to 30 mg m²/day for a 4-day course of clofarabine. Clofarabine will be started at Day -8 to allow improvement of liver function tests, if any, by time of allo-HSCT. Clofarabine (C) 30 mg/m²/day for 4 days (day -8 to day-5). Busilvex (B): 3.2 mg/kg/day for 2 days (day -4 and day-3)Thymoglobuline (T): 2.5 mg/Kg/day for 2 days (day -2 and day-1). Graft (G) at day 0 GVHD prophylaxis: Cyclosporine 3 mg/kg/day starting day-1. Genzyme provided supplies of clofarabine for all patients included in the study.

SUMMARY:
Clofarabine is known to have a stronger anti-tumor effect than Fludarabine and has shown its efficacy in treating aggressive acute leukemias. In addition, evidence is that it is well-tolerated with manageable side effects especially in elderly patients. Thus, replacing Fludarabine with Clofarabine in a reduced intensity transplant regimen may provide a regimen with increased anti-tumor activity without adding significant risks of toxicity.The purpose of this study is to evaluate the efficacy and the safety of clofarabine in combination with IV busulfan and ATG as the backbone of a reduced intensity conditioning regimen for allogeneic stem cell transplantation for the treatment of patients with high-risk MDS/AML or ALL not eligible to conventional or standard myeloablative allo-SCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* For patients younger than 50 years, cons-indication for the use of a standard myeloablative conditioning (history of hematopoietic stem cell transplantation autologous or allogeneic, or the presence of co-morbidities or medical history making prohibitive in terms toxicity using chemotherapy and / or high dose radiotherapy as judged by the referring physician) - MDS, ALL or AML at high risk, WHO THE biphenotypic-Score <2
* Any primary diagnosis of high-risk MDS/AML or ALL eligible for a treatment by reduced intensity conditioning (RIC) allogeneic hematopoietic stem cell transplantation (allo-SCT)
* Suitable donor available (related or matched unrelated)
* Cardiac: LV Ejection Fraction ≥ 50% by MUGA or Echocardiogram.
* Pulmonary: FEV1 and FVC ≥ 50% predicted, and DLCO (corrected for hemoglobin) ≥ 50% of predicted
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%
* Informed consent signed by patient prior to enrolment

Exclusion Criteria:

* Age <18
* Age >65
* Known hypersensitivity to clofarabine or excipients- Other hematologic malignancies than ALL, AML and MDS
* Patients with prior standard allogeneic HSCT with grade > 2 aGvHD
* Prior standard allogeneic transplantation if < 2 months
* Contra-indication to one of the drug of the RIC regimen .
* Patient with > 3 treatment lines prior to inclusion
* Pregnant or lactating females
* Patient HIV+, Hep B+, Hep C+- Uncontrolled systemic infection
* Performance Status Score ECOG > 2- Known central nervous system involvement with AML or ALL- Uncontrolled active infection of any kind or bleeding
* Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo the agents included in the conditioning regimen.
* For patients younger than 50 years, possibly indicating a standard myeloablative conditioning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relapse rate at one year after allo-SCT using the Clofarabine+Busulfan +Thymoglobuline reduced intensity conditioning regimen (CBT regimen). | at one year

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Nantes University hospital, Nantes
  - Hôpital Saint Louis, Paris
  - CHU Haut-Lévêque, Pessac
  - CHRU Hautepierre, Strasbourg

REFERENCES:
- [Derived] Chevallier P, Labopin M, Socie G, Tabrizi R, Furst S, Lioure B, Guillaume T, Delaunay J, de La Tour RP, Vigouroux S, El-Cheikh J, Blaise D, Michallet M, Bilger K, Milpied N, Moreau P, Mohty M. Results from a clofarabine-busulfan-containing, reduced-toxicity conditioning regimen prior to allogeneic stem cell transplantation: the phase 2 prospective CLORIC trial. Haematologica. 2014 Sep;99(9):1486-91. doi: 10.3324/haematol.2014.108563. Epub 2014 Jun 20. PMID 24951467